CLINICAL TRIAL: NCT03298477
Title: Prospective, Multicenter, Single Arm Safety and Effectiveness Confirmatory Study of Endovascular Abdominal Aortic Aneurysm Repair Using the Nellix System IDE Study (EVAS 2 Confirmatory IDE Study)
Brief Title: EVAS2 IDE Prospective, Multicenter, Single Arm Safety and Effectiveness Confirmatory Study
Acronym: EVAS2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0008 EVAS2 IDE
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single arm study with consecutive, eligible subject enrollment at each site. All subjects will undergo the Endovascular Aneurysm repair procedure with the Nellix System. Sites have been chosen with a suitable research infrastructure and physician experience in endovascular aneurysm repair to ensure adequate enrollment. Subjects will be followed procedurally to discharge, at 30 days (primary safety endpoint), six months, one year (primary effectiveness endpoint) and annually thereafter to five years (total follow-up commitment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Other): Single Arm Safety and Effectiveness Confirmatory Study of EVAS using the Nellix® System
  Interventions: Device: Nellix® System

INTERVENTIONS:
Device: Nellix® System — Endovascular Abdominal Aortic Aneurysm Repair using the Nellix® System

SUMMARY:
Prospective, multicenter, single arm study with consecutive, eligible subject enrollment at each site. All subjects will undergo the Endovascular Aneurysm repair procedure with the Nellix System.

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of the Nellix System among a wide range of physicians and in consecutively enrolled subjects to assess safety and effectiveness outcomes. Following appropriate government and ethics committee/IRB approval the Nellix® EndoVascular Sealing System will be implanted into eligible patients who are adequately informed and have consented to join the study. Enrolled patients will undergo a high resolution, contrast-enhanced computed tomography angiography (CT) scan of the relevant aortic and aortoiliac vasculature within three months of the scheduled procedure and at specified follow-up intervals post-implantation. Follow-up visits will occur at 30 days, 6 months, and annually to 5 years to assess aneurysm morphology, the status of the implanted devices, and relevant laboratory test results.

ELIGIBILITY:
INCLUSION CRITERIA

A patient who meets all of the following criteria potentially may be included in the study:

1. Male or female at least 18 years old;
2. Informed consent form understood and signed
3. Patient agrees to all follow-up visits;
4. Abdominal aortic aneurysm with sac diameter ≥5.0cm, or ≥4.5cm which has increased by ≥0.5cm within the last 6 months, or or which exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment. No AAA <4 cm will be included.
5. Anatomically eligible for the Nellix System (per Instructions For Use):

   1. Adequate iliac/femoral access compatible with the required delivery systems (diameter ≥6 mm);
   2. Aneurysm blood lumen diameter ≤60mm;
   3. Proximal non-aneurysmal aortic neck: length ≥10mm; diameter 18 to 28mm; angle ≤60° to the aneurysm sac;
   4. Most caudal renal artery to each hypogastric artery length ≥100mm;
   5. Common iliac artery lumen diameter between 9 and 35mm;
   6. Distal iliac artery seal zone with length of ≥10mm and diameter range of 9 to 25mm;
   7. Ability to preserve at least one hypogastric artery.
   8. Ratio of maximum aortic aneurysm diameter to maximum aortic blood lumen diameter <1.40

EXCLUSION CRITERIA

A patient who meets none of the following criteria potentially may be included in the study:

1. Life expectancy <2 years as judged by the Investigator;
2. Psychiatric or other condition that may interfere with the study;
3. Participating in another clinical study;
4. Known allergy or contraindication to any device material;
5. Coagulopathy or uncontrolled bleeding disorder;
6. Ruptured, leaking or mycotic aneurysm;
7. Serum creatinine (S-Cr) level >2.0 mg/dL;
8. CVA or MI within three months of enrollment/treatment;
9. Aneurysmal disease of the descending thoracic aorta;
10. Clinically significant mural thrombus within the proximal landing zone (minimum 10mm) of the infrarenal non-aneurysmal neck (>5mm thickness over >50% circumference);
11. Connective tissue diseases (e.g., Marfan Syndrome);
12. Unsuitable vascular anatomy that may interfere with device introduction or deployment;
13. Pregnant (female of childbearing potential only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2025-08-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Carpenter, MD, Principal Investigator — Cooper Hospital
Locations (27):
- United States (27):
  - Valley Vascular Consultants, Huntsville, Alabama
  - Regents of the University of California (UCLA), Los Angeles, California
  - Veterans Medical Research Foundation, San Diego, California
  - UC Health-Memorial Hospital, Colorado Springs, Colorado
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Miami Cardiac & Vascular Institute (MCVI), Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Coastal Vascular & Interventional, Pensacola, Florida
  - Christie Clinic, Champaign, Illinois
  - AMITA Health, Elk Grove Village, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - McLaren Bay Region, Bay City, Michigan
  - Midwest Aortic & Vascular Institute, Kansas City, Missouri
  - The Cooper Health System, Camden, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Northeast Ohio Vascular Assoc (NEOVA), Willoughby, Ohio
  - OU College of Medicine, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Palmetto Health- University of South Carolina, Columbia, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - Inova Research Center, Falls Church, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Aspirus Research Institute, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Nellix EndoVascular Aneurysm Sealing System: Nellix EndoVascular Aneurysm Sealing System: The study is designed to evaluate the safety, effectiveness and performance of the Nellix System for endovascular aneurysm repair. Subjects will be followed procedurally to discharge, at 30 days (primary safety endpoint), six months, one year, two year (primary effectiveness endpoint) and annually thereafter to five years (total follow-up commitment).
Period: 1 Month Follow-Up
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
Started | 98
Completed | 97
Not Completed | 1
Period: 6 Month Follow-Up
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
Started | 97
Completed | 93
Not Completed | 4
Period: 1 Year Follow-Up
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
Started | 93
Completed | 91
Not Completed | 2
Period: 2 Year Follow-Up
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
Started | 91
Completed | 81
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is 97 subjects. A total of 98 subjects were enrolled, with 97/98 subjects implanted with the Nellix System.
Groups:
- Single Arm Nellix EndoVascular Aneurysm Sealing System: All subjects will undergo the Endovascular Aneurysm repair procedure with the Nellix System. The study is designed to evaluate the safety, effectiveness and performance of the Nellix System for endovascular aneurysm repair. Subjects will be followed procedurally to discharge, at 30 days (primary safety endpoint), six months, one year, two years (primary effectiveness endpoint) and annually thereafter to five years (total follow-up commitment).
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 89
  Non Caucasian | 8
Region of Enrollment [Number; unit: participants]
  United States | 97
Height [Mean (Standard Deviation); unit: cm] | 177 (10)
ASA Class (ASA Physical Status Classification System) [Count of Participants; unit: Participants] — ASA 1: A normal healthy patient. No systemic disease. ASA 2: A patient with mild systemic disease. No significant impact on daily activity.
  ASA 3: A patient with severe systemic disease that limits activity but is not incapacitating. Significant impact on daily activity.
  ASA 4: A patient with severe systemic disease that is a constant threat to life. Life threatening conditions or multiple serious health issues.
  ASA 5: A moribund patient who is not expected to survive without the operation. Surgery is a last-ditch effort to save life.
  Participants
    ASA Class 1/2 | 32
    ASA Class 3/4/5 | 65
SVS Class (Society for Vascular Surgery Classification System) SVS/AAVS comorbidity score [Count of Participants; unit: Participants] — The overall SVS/AAVS comorbidity score is the sum of grades for the three organ systems (cardiac status, pulmonary status, and renal function):
  Low risk: Total score 0-3. Moderate risk: Total score 4-6. High risk: Total score 7-9.
  Participants
    SVS Score: 0/1 | 93
    SVS Score: 2/3/4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety: Major Adverse Events (MAE)
Description: The primary safety endpoint is defined as the incidence of Major Adverse Events (MAE) at 30 days, defined as the composite of the following All-Cause Mortality; Bowel Ischemia; Myocardial Infarction; Paraplegia; Renal Failure; Respiratory Failure; Stroke; Procedural Blood Loss ≥1,000cc
Time Frame: 30 days
Population: 98 patients enrolled under the study
Measure: Number; unit: Number of Events
Groups:
- Nellix System: Single Arm Safety and Effectiveness Confirmatory Study of EVAS using the Nellix® System
  Nellix® System: Endovascular Abdominal Aortic Aneurysm Repair using the Nellix® System
Arm/Group | Nellix System
Number analyzed (Participants) | 98
Number of Events
  Death | 1
  Myocardial Infarction | 2
  Renal Failure | 2

2. Primary Outcome: Effectiveness: Rate of Treatment Success
Description: The primary effectiveness endpoint is defined as the rate of Treatment Success at year 2. Treatment Success is a composite of outcomes clinically relevant to the endovascular repair of infrarenal AAA as follows:
  It is defined as procedural technical success and absence of Abdominal aortic aneurysm rupture; Conversion to open surgical repair; Endoleak Type I or III at year 2; Clinically significant migration; > 5mm aneurysm sac enlargement of the maximal diameter as measured by the difference from the 30-Day CT time point; or Secondary endovascular procedure up to year 2 for resolution of Endoleak (Type I or Type III), Device obstruction or occlusion, Device migration, Abdominal aneurysm sac expansion, Device defect.
Time Frame: 2 year
Population: Only 77 subjects completed study related procedures at 2 year time point.
Measure: Number; unit: percentage of treatment success
Arm/Group | Nellix System
Number analyzed (Participants) | 77
percentage of treatment success | 92.2

3. Secondary Outcome: Conversions, Death and Ruptures
Description: Number of Deaths, Conversion and ruptures through the data cut of the July 7, 2023,
Time Frame: 2 Years
Population: 93 subjects that completed their 2 year visit as of the data cut off of 07Jul2023
Measure: Number; unit: Number of Events
Groups:
- Nellix EndoVascular Aneurysm Sealing System: Nellix EndoVascular Aneurysm Sealing System: The System is designed to evaluate the safety and Effectiveness and performance of the Nellix System for endovascular aneurysm repair in subjects implanted with it. Subjects will be followed procedurally to discharge, at 30 days (primary safety endpoint), six months, one year, two year (primary effectiveness endpoint) and annually thereafter to five years (total follow-up commitment).
Arm/Group | Nellix EndoVascular Aneurysm Sealing System
Number analyzed (Participants) | 93
Number of Events
  Conversion | 0
  Deaths | 7
  Ruptures | 0

4. Secondary Outcome: Device Integrity
Description: Device Integrity is defined as the absence of device fracture, stenosis, kink, occlusion, or migration >5mm. All incidences of stent occlusion (100% device lumen obstruction) are also captured as stent stenosis (<100% device lumen obstruction).
Time Frame: 2 Years
Population: 75 participants that were analyzed for device integrity as of 07Jul2023, Data for >5mm Migration includes subjects with Migration >10mm as well.
Measure: Number; unit: Number of Events
Groups:
- Nellix EndoVascular Aneurysm Sealing System:: Nellix EndoVascular Aneurysm Sealing System: The System is designed to evaluate the safety and Effectiveness and performance of the Nellix System for endovascular aneurysm repair in subjects implanted with it. Subjects will be followed procedurally to discharge, at 30 days (primary safety endpoint), six months, one year, two year (primary effectiveness endpoint) and annually thereafter to five years (total follow-up commitment).
Arm/Group | Nellix EndoVascular Aneurysm Sealing System:
Number analyzed (Participants) | 75
Number of Events
  Stenosis | 5
  Stent Occlusion | 4
  Migration>5mm | 1
  Migration >10mm | 0
  Stent Kinking | 0
  Stent Fracture | 0

5. Secondary Outcome: Device Performance - Endoleak
Description: Demonstrates device performance as indicated by the incidence of Endoleaks through study follow-up. Endoleak is determined by the CoreLab based on imaging completed. Endoleak is defined as clear evidence of contrast outside of one or both EndoBags which communicates with the aneurysm sac originating proximally at the infrarenal segment (Type IA), distally (Type IB); between components, if an extender is used (Type III); trans-device (Type IV); or from a patent collateral vessel (Type II: e.g., lumbar artery; inferior mesenteric artery).
Time Frame: 2 Years
Population: 75 subjects analyzed for Endoleaks at 2 years as of the data cut-off date of 07Jul2023
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm Nellix EndoVascular Aneurysm Sealing System: Nellix® System: Endovascular Abdominal Aortic Aneurysm Repair using the Nellix® System
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
Number analyzed (Participants) | 75
Participants
  Endoleak Type IA | 5
  Endoleak Type IB | 1
  Endoleak Type II | 6
  Endoleak Type III | 0
  Endoleak Type IV | 0
  Endoleak Unknown | 1

6. Secondary Outcome: DEVICE PERFORMANCE-ANEURYSM SAC DIAMETER- Avg Size
Description: Average Sac Diameter size at Visit
Time Frame: 2 years
Population: 76 Subjects that were analyzed at 2 years for Average Sac size in diameters as of the data cut-off date of 07Jul2023
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Nellix System
Number analyzed (Participants) | 76
mm | 55.4 (5.9)

7. Secondary Outcome: DEVICE PERFORMANCE-ANEURYSM SAC DIAMETER- Changes in Sac Size Since 01 Month
Description: Number of subjects that had changes in the Sac Diameter size since the 1 month follow-up visit
Time Frame: 2 Years
Population: 76 Subjects that were analyzed at 2 years for changes in Diameter sac Changes since 1month as of the cutoff date of 07Jul2023
Measure: Number; unit: Number of subjects
Arm/Group | Nellix System
Number analyzed (Participants) | 76
Number of subjects
  Decreased >5mm | 3
  Stable +- 5mm | 69
  Increased >5mm | 4
  No Growth | 72

8. Secondary Outcome: Secondary Interventions
Description: All Secondary interventions reported during the study
Time Frame: 2 Years
Population: 93 subjects analyzed for the number of secondary interventions
Measure: Number; unit: Number of Events
Arm/Group | Nellix System
Number analyzed (Participants) | 93
Number of Events
  Conversion to open repair due to aneurysm expansion | 0
  Iliac Extension due to aneurysm expansion | 1
  Iliac Stenting due to renal failure | 1
  Renal stent due to renal failure | 1
  Iliac Extension due to Vessel Dissection (Non aortic) | 1
  Thrombolysis due to Vessel Dissection (Non aortic) | 1
  Conversion to Open Repair due to endoleak IA | 0
  Coil Embolization due to Endoleak II | 1
  Thrombolysis due to Stent Thrombosis | 2
  Stent relining due to Stent Thrombosis | 1
  Fem-Fem Bypass due to Stent Thrombosis | 1
  Conversion to Open Repair due to stent migration | 0
  Renal stent due to Renal Artery Occlusion | 1

9. Secondary Outcome: LABS-RENAL FUNCTION (EGFR)
Description: The outcome demonstrates the protocol specified laboratory values (collected as eGFR) captured at each follow-up visit
Time Frame: 2 Years
Population: 80 subjects analyzed for renal function (eGFR) at 2 years as of the data cut-off date of 07Jul2023
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Nellix System
Number analyzed (Participants) | 80
mL/min/1.73 m^2 | 66 (24)

10. Secondary Outcome: LABS- RENAL FUNCTION (CREATININE)
Description: Labs- Renal Function demonstrates the protocol specified laboratory values (Collected as creatinine) captured at each follow-up visit
Time Frame: 2 Years
Population: 80 subjects analyzed for renal function (Creatinine) at 2 years as of the data cut-off date of 07Jul2023
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nellix System
Number analyzed (Participants) | 80
mg/dL | 1.19 (0.42)

ADVERSE EVENTS:
Time Frame: All Adverse Events data occurring during the study period were collected (i.e. procedure through 5 years follow-up). The data reported here are as of the data cut for 2-year primary endpoint data.
Arm/Group | Single Arm Nellix EndoVascular Aneurysm Sealing System
All-Cause Mortality (participants affected / at risk) | 7/98
Serious Adverse Events (participants affected / at risk) | 49/98
Other Adverse Events (participants affected / at risk) | 22/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Nellix EndoVascular Aneurysm Sealing System (N=98)
Bleeding/Anemia (Blood and lymphatic system disorders) | 5 (5)
Bowel (Gastrointestinal disorders) | 4 (4)
Cardiac (Cardiac disorders) | 11 (13)
Chimney Device (Surgical and medical procedures) | 0 (0)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Miscellaneous (General disorders) | 19 (20)
Nellix Device (Product Issues) | 4 (6)
Neurological (Nervous system disorders) | 5 (5)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Renal (Renal and urinary disorders) | 8 (8)
Surgical Site Wound (Surgical and medical procedures) | 1 (1)
Urogenital (Renal and urinary disorders) | 5 (5)
Vascular (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Nellix EndoVascular Aneurysm Sealing System (N=98)
Bleeding/Anemia (Blood and lymphatic system disorders) | 0 (0)
Bowel (Gastrointestinal disorders) | 1 (1)
Cardiac (Cardiac disorders) | 3 (3)
Nellix Device (Product Issues) | 1 (1)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Miscellaneous (General disorders) | 12 (15)
Chimney Device (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Neurological (Nervous system disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Renal (Renal and urinary disorders) | 3 (3)
Surgical Site Wound (Surgical and medical procedures) | 1 (1)
Urogenital (Renal and urinary disorders) | 5 (5)
Vascular (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT03298477/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03298477/ICF_001.pdf